CLINICAL TRIAL: NCT02935491
Title: 4 Cities for Assessing CAlcification PRognostic Impact After TAVI
Acronym: C4CAPRI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0651
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Heart Disease
Keywords: TAVI; Aortic stenosis; aortic stiffness; calcifications; CT-scan; Vascular impedance
MeSH Terms: conditions — Heart Diseases; Aortic Valve Stenosis; Calcinosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transcatheter Aortic Valve Implantation: Lyon and Paris cohorts : 900 patients will be used to test the prognostic value of aortic calcifications and to propose a risk score Clermont and Rouen cohorts (700 patients) will be used to test in an independent group, the predictive value of the risk score
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — TAVI is a well-accepted method for aortic valve replacement without surgery. It is currently proposed to patients at high surgical risk or contraindicated to surgery. It consists of introducing a valve inserted inside a stent by the femoral artery in most cases.
  Aortic calcifications will be determined by the analysis of the CT-scan performed systematically before the procedure. A semi-automated software (CreaTools) will be used

SUMMARY:
Transcatheter Aortic Valve Implantation (TAVI) indications are progressing rapidly as an alternative to conventional surgery for aortic stenosis cure. Despite a high rate of procedural success, some patients do not benefit from the procedure. The investigators hypothesis is that aortic stiffness may be of major prognostic significance after stenosis relief.

The aim of this study is to test the prognostic impact of aortic stiffness estimated by the volume of calcifications of the thoracic aorta on the CT-scan performed systematically before the procedure. This prognostic value will be assessed in 4 independent cohorts issued from 4 french cities (Lyon, Rouen, Paris, Clermont-Ferrand).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patient who underwent a transcatheter aortic valve implantation
* Patient who provided informed, written consent to participate to FRANCE TAVI study
* Patient for whom a CT-Scan performed before TAVI procedure is available.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sex presenting with a severe aortic stenosis with the indication of aortic replacement by TAVI
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | censored on 3 March 2017
  Number of death of cardiovascular cause will be analyzed

SECONDARY OUTCOMES:
All-cause deaths | censored on 3 March 2017
  Number of death of all causes will be analyzed
left ventricular remodeling | censored on 3 March 2017
  Echocardiographic measure will be done
left ventricular ejection fraction | censored on 3 March 2017
  Echocardiographic measure will be done
diastolic function | censored on 3 March 2017
  Echocardiographic measure will be done

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France